CLINICAL TRIAL: NCT01102218
Title: A Randomized Multi-Center Study to Determine the Safety and Efficacy of Erythropoietin Plus Pentoxifylline Versus Erythropoietin Alone for the Treatment of Anemia in Subjects With End Stage Renal Disease on Maintenance Hemodialysis
Brief Title: A Safety Study of Pentoxifylline for the Treatment of Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of statistical difference between both arms of the trial.
Sponsor: Fresenius Medical Care North America (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-01
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: End Stage Renal Disease
Keywords: Anemia, ESRD
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia | interventions — Erythropoietin; Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- erythropoietin plus pentoxifylline (Experimental)
  Interventions: Drug: Erythropoietin; Drug: Pentoxifylline
- erythropoietin alone (Active Comparator)
  Interventions: Drug: Erythropoietin

INTERVENTIONS:
Drug: Erythropoietin — Standard of Care
  Arms: erythropoietin plus pentoxifylline
Drug: Erythropoietin — Standard of Care
  Arms: erythropoietin alone
Drug: Pentoxifylline — 400 mg qd po for 6 months
  Other Names: brand name is Trental
  Arms: erythropoietin plus pentoxifylline

SUMMARY:
Chronic kidney disease (CKD) patients have increased levels of inflammation and oxidative stress, which in turn contribute to anemia and cardiovascular disease.

Pentoxifylline is known to have anti-inflammatory and anti-oxidant properties, and has shown promise in improving the treatment of patients with anemia. This study will examine the use of pentoxifylline for the treatment of anemia in chronic kidney disease.

DETAILED DESCRIPTION:
Treatment of the anemia of renal failure has been revolutionized by the use of erythropoietin and other ESAs (erythropoiesis-stimulating agent). Concerns with ESA use include a substantial number of End Stage Renal Disease (ESRD) patients with ESA-resistant anemia, and a growing body of evidence of potential negative effects of high doses of ESA use, including increased mortality and increased rate of tumor growth in cancer patients.

There are only a couple of small studies in the literature examining the effects of pentoxifylline on anemia in patients with renal failure. The results are limited by the very small number of patients. There is clearly a need for a larger, prospective, clinical trial of pentoxifylline in ESRD patients, not limited to those with ESA-resistant anemia. This would be the first prospective, randomized clinical trial of this size to study pentoxifylline for the treatment of anemia in chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥18 years;
* Able to comply with the study procedures and medication;
* Written informed consent given;
* On a stable in-center hemodialysis regimen (at least 3 times per week) for ≥ 12 weeks prior to screening;
* Subject must have been on a stable (< 25% change) erythropoietin dose with an average of ≥ 15,000 and <55,000 units/week of treatment for ≥ 14 days prior to screening visit;
* Two hemoglobin measurements must meet the following criteria: (1) Taken ≥ 2 weeks apart; (2) Between 10 and 12 g/dL, inclusive; (3) Within 1 g/dL of each other; and (4) Occurred within 30 days prior to screening visit;
* If subject is a female and of childbearing potential (pre-menopausal and not surgically sterile), subject is willing to use an effective contraceptive method throughout study, which includes abstinence, barrier methods, hormones, or IUDs;
* Life expectancy of 12 months or greater;
* Most recent single pool Kt/V ≥1.2, taken within 45 days prior to screening visit;
* Stable nutrition status with all albumin levels ≥ 3.0 g/dL within the 30 days prior to screening visit.

Exclusion Criteria:

* Participation in any clinical trial using an investigational product or device during the 30 days preceding the Screening Visit;
* Currently undergoing nocturnal hemodialysis;
* A significant history of alcohol, drug or solvent abuse in the opinion of the investigator;
* Serum iPTH > 800 pg/mL within 90 days prior to screening visit;
* Dysrhythmia or severe cardiac disease: CHF Class III-IV; unstable cardiovascular diagnosis (for example MI, CABG, PTCA, CVA, and TIA) within 90 days prior to screening visit;
* Significant concurrent liver disorder [Aspartate transaminase (AST) or alanine transaminase (ALT) values > 3 times upper limit of normal (ULN) within 30 days prior to screening];
* Platelet count < 130x109 within 30 days prior to screening visit or on the day of the screening visit;
* Known hypersensitivity to, or intolerance of, Pentoxifylline or other methylxanthines, such as caffeine, theophylline or theobromine;
* Currently taking pentoxifylline, warfarin, theophylline, aminophylline, dyphylline, or oxtriphylline;
* Absolute or functional iron deficiency [transferrin saturation (TSAT) <20%] within 45 days prior to screening;
* Recent or severe hemorrhage per PI discretion;
* Significant bleeding episode or prolonged bleeding from dialysis access per PI judgment within the 3 months prior to screening;
* Melatonin treatment, androgen therapy or blood transfusion within 30 days prior to screening;
* Vitamin C therapy at dose greater than 100 mg/day or at a dose which has changed within the last 3 months;
* Current active cancer (excluding basal cell carcinoma of the skin);
* Poorly controlled hypertension per PI judgment within 4 weeks prior to screening;
* Known HIV positive status;
* Significant GI disorders where absorption of an oral medication might, in the opinion of the Investigator, be impaired;
* Anticipated live donor kidney transplant or any other planned major surgery over the study duration;
* History of poor adherence to hemodialysis or medical regimen;
* Any active clinically significant infection or evidence of an underlying infection;
* Currently on immunosuppressive drug regimen other than a stable, low dose of steroids, per PI judgment;
* Any disease or condition, physical or psychological that, in the opinion of the investigator, would compromise the safety of the subject or the likelihood of achieving reliable results or increase the likelihood of the subject being withdrawn.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond M. Hakim, MD, PhD, Principal Investigator — Fresenius Medical Care North America
Locations (10):
- United States (10):
  - Fresenius Medical Care North America, Chicago, Illinois
  - Fresenius Medical Care North America, Kalamazoo, Michigan
  - Fresenius Medical Care North America, Brookhaven, Mississippi
  - Fresenius Medical Care North America, Tupelo, Mississippi
  - Fresenius Medical Care North America, City of Saint Peters, Missouri
  - Fresenius Medical Care North America, Saint Ann, Missouri
  - Fresenius Medical Care North America, Las Vegas, Nevada
  - Fresenius Medical Care North America, Columbia, Tennessee
  - Fresenius Medical Care North America, Irving, Texas
  - Fresenius Medical Care North America, Tyler, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Fresenius Medical Care North America Dialysis clinics between August 2010 and October 2011.
Pre-assignment Details: There was no wash out or run in period for this trial.68 subjects signed informed consent, and 48 subjects were randomized.13 of the 20 screen failures were due to exclusionary lab values, 3 due to excluded medications, and 3 were due to other exclusion criteria, 1 due to unrelated SAE. Zero patients withdrew consent prior to randomization.
Groups:
- Erythropoietin Plus Pentoxifylline: Standard of care prescribed erythropoietin dose plus 400mg oral pentoxifylline once a day.
- Erythropoietin Alone: Standard of care prescribed erythropoietin dose.
Period: Overall Study
Arm/Group | Erythropoietin Plus Pentoxifylline | Erythropoietin Alone
Started | 24 | 24
Completed | 13 | 14
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Erythropoietin Plus Pentoxifylline | Erythropoietin Alone | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 35
  >=65 years | 5 | 8 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (12) | 57 (14) | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Erythropoietin Dose
Description: Erythropoietin dose is amount needed to maintain a hemoglobin between 11 and 12 mg/dL.
Time Frame: Baseline and 6 months
Population: The number of patients for analysis was based on those patient who had completed 6 months of treatment. The analysis was per protocol.
Measure: Mean (Standard Deviation); unit: Units EPO
Arm/Group | Erythropoietin Plus Pentoxifylline | Erythropoietin Alone
Number analyzed (Participants) | 9 | 8
Units EPO | -8700 (12586) | -2988 (10232)
Statistical Analysis 1: Comparison: Erythropoietin Plus Pentoxifylline vs Erythropoietin Alone; Test type: Superiority or Other; p > 0.05, ANCOVA

2. Secondary Outcome: Examine the EPO Resistance Index (Erythropoietin Dose/kg/Week/Hgb) or ERI Over Time
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Observe Changes in Markers of Inflammation Including But Not Limited to TNF-α and IL-6
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Erythropoietin Plus Pentoxifylline | Erythropoietin Alone
Serious Adverse Events (participants affected / at risk) | 12/24 | 12/24
Other Adverse Events (participants affected / at risk) | 22/24 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin Plus Pentoxifylline (N=24) | Erythropoietin Alone (N=24)
Infection (Infections and infestations) | 2 (3) | 3 (5)
Cardiac (Cardiac disorders) | 5 (5) | 1 (1)
Access related (Vascular disorders) | 1 (2) | 2 (2)
Dizziness (General disorders) | 0 (0) | 2 (2)
Fluid overload (Cardiac disorders) | 1 (2) | 0 (0)
Other (General disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diabetes (Endocrine disorders) | 0 (0) | 1 (1)
Electrolyte disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GI upset (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erythropoietin Plus Pentoxifylline (N=24) | Erythropoietin Alone (N=24)
GI upset (Gastrointestinal disorders) | 6 (13) | 6 (11)
Infection (Infections and infestations) | 5 (6) | 7 (13)
Access-related (Vascular disorders) | 3 (7) | 4 (6)
Other (General disorders) | 2 (5) | 3 (3)
Pain (General disorders) | 4 (5) | 2 (2)
Cardiac (Cardiac disorders) | 2 (2) | 2 (3)

LIMITATIONS AND CAVEATS:
Release of new FDA guidelines re target Hgb values impacted EPO dosing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After Sponsor's (S) publication (pub) of multi-center pub,Institution (I) and/or Principal Investigator (PI) may publish data/results from Study based solely upon Study conducted by I/PI,provided that I/PI submits pub to S for review/comment > 60 days before date of proposed pub.S may review in advance contents of pub.If pub is not submitted within 12 months after termination of Study at all sites,or if S confirms there will be no pub,the I/PI may publish Study results.